CLINICAL TRIAL: NCT03007524
Title: A Randomized Comparison of Low-dose Versus High-dose Rosuvastatin on Optical Coherence Tomography Based Early Vascular Healing for Patients With Acute Coronary Syndrome
Brief Title: Early Vascular Healing in Acute Coronary Syndrome Patients With Different Doses of Rosuvastatin
Acronym: CROWN-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yao-Jun Zhang, Principal Investigator, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20160608-02
Record Dates: First submitted 2016-07-12; First posted 2017-01-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Acute Coronary Syndrome
Keywords: rosuvastatin; optical coherence tomography; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose rosuvastatin (Experimental): 20mg/d quaque nocte(qN), at least 6 months
  Interventions: Drug: High dose Rosuvastatin
- Low dose rosuvastatin (Active Comparator): 10mg/d quaque nocte（qN）, at least 6 months
  Interventions: Drug: Low dose Rosuvastatin

INTERVENTIONS:
Drug: High dose Rosuvastatin — 20mg/d qN, at least 6 months
  Other Names: Rosuvastatin Calcium; Crestor
  Arms: High dose rosuvastatin
Drug: Low dose Rosuvastatin — 10mg/d qN, at least 6 months
  Other Names: Rosuvastatin Calcium; Crestor
  Arms: Low dose rosuvastatin

SUMMARY:
This is a prospective, randomized trial comparing different doses of rosuvastatin in patients with acute coronary syndrome post drug-eluting stents implantation. Through the study, the investigators aim to evaluate the effects of high dose rosuvastatin calcium on "target vessel" endothelialization and "non-target vessel" plaque stability. Moreover, the investigators may provide mechanically evidence of clinical application of high dose rosuvastatin in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled clinical trial comparing different doses of rosuvastatin in patients with acute coronary syndrome post drug-eluting stents implantation. In total, the investigators plan to recruit 80 patients with acute coronary syndrome (but no acute ST-segment elevation myocardial infarction) participating in the study. After signing informed consent form, the patients will be randomly assigned into high dose rosuvastatin and low dose rosuvastatin groups (40 cases in each group) by a computer generated random sequence table on a ratio of 1:1. Patients in the high-dose group will be prescribed rosuvastatin calcium of 20mg/d at least 6 months post index procedure, while patients in low dose group will have rosuvastatin calcium of 10mg/d, also at least 6 months. Additionally, all patients will receive dual antiplatelet therapy (oral aspirin 100mg qd, clopidogrel 75mg qd or ticagrelor 90 mg bid). Clinical follow up (telephone or out-patient follow-up) will be scheduled at 30 days, 6 months, 1 year, 2 years and 3 years. Optical coherence tomography examinations will be performed at 6 months. Neointimal hyperplasia, stent strut coverage and thin cap fibroatheroma are primary observational parameters. Multi-slices CT are optional pre-/post-procedure and at 3 years follow-up. All clinical data will be collected and managed by statistical center, clinical endpoint adjudication committee. All imaging modalities data will be collected and analysed by an independent imaging core laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years male or non-pregnant female;
2. Clinical evidence of unstable angina or non ST segment elevation myocardial infarction (NSTEMI);
3. The patient has up to two de novo native coronary lesions in different epicardial vessels;
4. Target lesion diameter stenosis ≧70%(visually estimated);
5. Each target lesion must be treated with maximal 2 stents (except the bailout stenting);
6. Low density lipoprotein (LDL) higher than 100mg/dL or lower than 100mg/dL but have taken statin drugs less than 1 month before enrolled;
7. Patient is an acceptable candidate for emergency coronary artery bypass grafting;
8. The patient is able to understand the aim of this study, provide voluntarily written informed content and agree to the follow-up visits including angiographic、multislice spiral computed tomography(MSCT) and optical coherence tomography(OCT) examinations;

Exclusion Criteria:

1. Any acute myocardial infarction within the past 1 months; myocardial enzyme not back to normal after myocardial infarction;
2. Chronic total occlusive lesion, severe left main coronary artery disease, orifice lesion, 3-vessel disease, bifurcation lesions (with side branch diameter greater than 2 mm, orifice diameter stenosis greater than or equal to 50%, or side branch need to be protected by guidewire or balloon), OCT imaging is not suitable for the lesion site or OCT imaging is incomplete, Target lesion located in previous venous or arterial bypass grafts, Target lesion has visible thrombus, intercurrent infection, or other inflammatory diseases.;
3. Heavily calcified lesions, severely tortuous lesions, lesions cannot be well pre-dilated and/or unsuitable of the stent crossover/expansion;
4. In-stent restenosis lesions;
5. Prior percutaneous coronary intervention(PCI) within the past 1 year; plan to possibly have re-intervention within 1 year post index-procedure; previous PCI more than 1 year at the target vessel;
6. Instability of hemodynamic or respiratory cycle, such as cardiogenic shock, Heart failure with severe symptoms (over New York Heart Association III(NYHA III)) or left ventricular ejection fraction less than 40% (UCG or left ventricle radiography);
7. Known renal insufficiency (e.g, Glomerular filtration rate(eGFR) <60 ml/kg/m2 or serum creatinine level of >2.5 mg/dL, or subject on dialysis);
8. History of bleeding tendency, active peptic ulcer and cerebral hemorrhage or retinal hemorrhage, and a half years history of stroke, antiplatelet agents and anticoagulants therapy contraindications to anticoagulation in patients;
9. Patients have been used statins and other lipid-lowering drug treatment more than 1 month before enrolled,patients allergy to rosuvastatin or use rosuvastatin with contraindications,patients allergy to aspirin, clopidogrel or ticagrelor, heparin, contrast agent, polymer, zotarolimus and metal;
10. Life expectancy <6 months;
11. Currently participating in an investigational drug or another device study that has not completed the primary endpoint;
12. Unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements;
13. The patient is a recipient of a heart transplant;
14. Unstable arrhythmia, such as high risk ventricular contraction, ventricular arrhythmia;
15. With the need of chemotherapy in 30 days due to malignancy;
16. Patients with immune suppression or autoimmune diseases planning to have or currently receive immunosuppressive therapy;
17. Patients planning to have or currently receive long-term anticoagulation therapy;
18. Patients may receive surgery within 6 months post index-procedure in which needs to stop aspirin, clopidogrel or ticagrelor;
19. Neutropenia (<1000 neutrophils/mm3), Thrombocytopenia (<100,000 platelets/mm3), Confirmed or suspected diagnosis of liver diseases;
20. Patients with diffuse peripheral vascular disease which precludes 6 French unit(6F) sheath insertion;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of covered struts | 6 months

SECONDARY OUTCOMES:
Mean/Minimal stent diameter | 6 months
Mean/Minimal stent area | 6 months
Mean/Minimal stent volume | 6 months
Mean/Minimal lumen diameter | 6 months
Mean/Minimal lumen area | 6 months
Mean/Minimal lumen volume | 6 months
Mean/Minimal vessel diameter | 6 months
Mean/Minimal vessel area | 6 months
Mean/Minimal vessel volume | 6 months
Mean/Minimal thickness of stent strut coverage | 6 months
thin cap fibroatheroma(TCFA) | 6 months
Cap thickness of thin cap fibroatheroma(TCFA) | 6 months
Neointimal Hyperplasia area | 6 months
Neointimal Hyperplasia volume | 6 months
Incomplete strut apposition | 6 months
Device-oriented composite endpoint | 1 and 6 months, 1, 2, 3 years
Cardiac death | 1 and 6 months, 1, 2, 3 years
Non-fatal myocardial infarction | 1 and 6 months, 1, 2, 3 years
All revascularization | 1 and 6 months, 1, 2, 3 years
target lesion revascularization | 1 and 6 months, 1, 2, 3 years
target vessel revascularization | 1 and 6 months, 1, 2, 3 years
stent thrombosis | 1 and 6 months, 1, 2, 3 years

OTHER OUTCOMES:
Lipid levels | Baseline，6 months
  Total cholesterol（TC）,low density lipoprotein(LDL),high density lipoprotein(HDL),LDL/HDL,triglyceride
Biological index | Baseline，6 months
  High sensitivity c-reactive protein（hs-CRP）,Pentraxin-3(PTX-3),Vascular cell adhesion molecule-1(VCAM-1),Matrix metallopeptidase-9(MMP-9)

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Jun Zhang, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Ze-Ning Jin, PhD, Principal Investigator — Beijing Anzhen Hospital; Fei Ye, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Song Lin, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Bo Xu, MSc, Study Director — Fu Wai Hospital, Beijing, China
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morice MC, Serruys PW, Barragan P, Bode C, Van Es GA, Stoll HP, Snead D, Mauri L, Cutlip DE, Sousa E. Long-term clinical outcomes with sirolimus-eluting coronary stents: five-year results of the RAVEL trial. J Am Coll Cardiol. 2007 Oct 2;50(14):1299-304. doi: 10.1016/j.jacc.2007.06.029. Epub 2007 Sep 17. PMID 17903626
- [Background] Grech ED. ABC of interventional cardiology: percutaneous coronary intervention. I: history and development. BMJ. 2003 May 17;326(7398):1080-2. doi: 10.1136/bmj.326.7398.1080. No abstract available. PMID 12750213
- [Background] Gottsauner-Wolf M, Zasmeta G, Hornykewycz S, Nikfardjam M, Stepan E, Wexberg P, Zorn G, Glogar D, Probst P, Maurer G, Huber K. Plasma levels of C-reactive protein after coronary stent implantation. Eur Heart J. 2000 Jul;21(14):1152-8. doi: 10.1053/euhj.1999.1987. PMID 10924298
- [Background] Walter DH, Fichtlscherer S, Britten MB, Rosin P, Auch-Schwelk W, Schachinger V, Zeiher AM. Statin therapy, inflammation and recurrent coronary events in patients following coronary stent implantation. J Am Coll Cardiol. 2001 Dec;38(7):2006-12. doi: 10.1016/s0735-1097(01)01662-x. PMID 11738308
- [Background] Losordo DW, Isner JM, Diaz-Sandoval LJ. Endothelial recovery: the next target in restenosis prevention. Circulation. 2003 Jun 3;107(21):2635-7. doi: 10.1161/01.CIR.0000071083.31270.C3. No abstract available. PMID 12782613
- [Background] Komatsu R, Ueda M, Naruko T, Kojima A, Becker AE. Neointimal tissue response at sites of coronary stenting in humans: macroscopic, histological, and immunohistochemical analyses. Circulation. 1998 Jul 21;98(3):224-33. doi: 10.1161/01.cir.98.3.224. PMID 9697822
- [Background] Mora S, Glynn RJ, Hsia J, MacFadyen JG, Genest J, Ridker PM. Statins for the primary prevention of cardiovascular events in women with elevated high-sensitivity C-reactive protein or dyslipidemia: results from the Justification for the Use of Statins in Prevention: An Intervention Trial Evaluating Rosuvastatin (JUPITER) and meta-analysis of women from primary prevention trials. Circulation. 2010 Mar 9;121(9):1069-77. doi: 10.1161/CIRCULATIONAHA.109.906479. Epub 2010 Feb 22. PMID 20176986
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Kearney PM, Blackwell L, Collins R, Keech A, Simes J, Peto R, Armitage J, Baigent C. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a meta-analysis. Lancet. 2008 Jan 12;371(9607):117-25. doi: 10.1016/S0140-6736(08)60104-X. PMID 18191683
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Mihaylova B, Emberson J, Blackwell L, Keech A, Simes J, Barnes EH, Voysey M, Gray A, Collins R, Baigent C. The effects of lowering LDL cholesterol with statin therapy in people at low risk of vascular disease: meta-analysis of individual data from 27 randomised trials. Lancet. 2012 Aug 11;380(9841):581-90. doi: 10.1016/S0140-6736(12)60367-5. Epub 2012 May 17. PMID 22607822
- [Background] Brugts JJ, Yetgin T, Hoeks SE, Gotto AM, Shepherd J, Westendorp RG, de Craen AJ, Knopp RH, Nakamura H, Ridker P, van Domburg R, Deckers JW. The benefits of statins in people without established cardiovascular disease but with cardiovascular risk factors: meta-analysis of randomised controlled trials. BMJ. 2009 Jun 30;338:b2376. doi: 10.1136/bmj.b2376. PMID 19567909
- [Background] Hou W, Lv J, Perkovic V, Yang L, Zhao N, Jardine MJ, Cass A, Zhang H, Wang H. Effect of statin therapy on cardiovascular and renal outcomes in patients with chronic kidney disease: a systematic review and meta-analysis. Eur Heart J. 2013 Jun;34(24):1807-17. doi: 10.1093/eurheartj/eht065. Epub 2013 Mar 6. PMID 23470492
- [Background] Ray KK, Cannon CP, Ganz P. Beyond lipid lowering: What have we learned about the benefits of statins from the acute coronary syndromes trials? Am J Cardiol. 2006 Dec 4;98(11A):18P-25P. doi: 10.1016/j.amjcard.2006.09.016. Epub 2006 Sep 29. PMID 17126675
- [Background] Almuti K, Rimawi R, Spevack D, Ostfeld RJ. Effects of statins beyond lipid lowering: potential for clinical benefits. Int J Cardiol. 2006 Apr 28;109(1):7-15. doi: 10.1016/j.ijcard.2005.05.056. Epub 2005 Jul 28. PMID 16054715
- [Background] Liu T, Li L, Korantzopoulos P, Liu E, Li G. Statin use and development of atrial fibrillation: a systematic review and meta-analysis of randomized clinical trials and observational studies. Int J Cardiol. 2008 May 23;126(2):160-70. doi: 10.1016/j.ijcard.2007.07.137. Epub 2007 Nov 26. PMID 18031847
- [Background] Marui N, Offermann MK, Swerlick R, Kunsch C, Rosen CA, Ahmad M, Alexander RW, Medford RM. Vascular cell adhesion molecule-1 (VCAM-1) gene transcription and expression are regulated through an antioxidant-sensitive mechanism in human vascular endothelial cells. J Clin Invest. 1993 Oct;92(4):1866-74. doi: 10.1172/JCI116778. PMID 7691889
- [Background] Karalis IK, Bergheanu SC, Wolterbeek R, Dallinga-Thie GM, Hattori H, van Tol A, Liem AH, Wouter Jukema J. Effect of increasing doses of Rosuvastatin and Atorvastatin on apolipoproteins, enzymes and lipid transfer proteins involved in lipoprotein metabolism and inflammatory parameters. Curr Med Res Opin. 2010 Oct;26(10):2301-13. doi: 10.1185/03007995.2010.509264. PMID 20731529
- [Background] Kleemann R, Princen HM, Emeis JJ, Jukema JW, Fontijn RD, Horrevoets AJ, Kooistra T, Havekes LM. Rosuvastatin reduces atherosclerosis development beyond and independent of its plasma cholesterol-lowering effect in APOE*3-Leiden transgenic mice: evidence for antiinflammatory effects of rosuvastatin. Circulation. 2003 Sep 16;108(11):1368-74. doi: 10.1161/01.CIR.0000086460.55494.AF. Epub 2003 Aug 25. PMID 12939225
- [Background] Llevadot J, Murasawa S, Kureishi Y, Uchida S, Masuda H, Kawamoto A, Walsh K, Isner JM, Asahara T. HMG-CoA reductase inhibitor mobilizes bone marrow--derived endothelial progenitor cells. J Clin Invest. 2001 Aug;108(3):399-405. doi: 10.1172/JCI13131. PMID 11489933
- [Background] Weber C, Erl W, Weber KS, Weber PC. HMG-CoA reductase inhibitors decrease CD11b expression and CD11b-dependent adhesion of monocytes to endothelium and reduce increased adhesiveness of monocytes isolated from patients with hypercholesterolemia. J Am Coll Cardiol. 1997 Nov 1;30(5):1212-7. doi: 10.1016/s0735-1097(97)00324-0. PMID 9350917
- [Background] Mizukoshi M, Imanishi T, Tanaka A, Kubo T, Liu Y, Takarada S, Kitabata H, Tanimoto T, Komukai K, Ishibashi K, Akasaka T. Clinical classification and plaque morphology determined by optical coherence tomography in unstable angina pectoris. Am J Cardiol. 2010 Aug 1;106(3):323-8. doi: 10.1016/j.amjcard.2010.03.027. PMID 20643240
- [Background] Akasaka T, Kubo T, Mizukoshi M, Tanaka A, Kitabata H, Tanimoto T, Imanishi T. Pathophysiology of acute coronary syndrome assessed by optical coherence tomography. J Cardiol. 2010 Jul;56(1):8-14. doi: 10.1016/j.jjcc.2010.05.005. Epub 2010 Jun 15. PMID 20554431
- [Background] Bezerra HG, Costa MA, Guagliumi G, Rollins AM, Simon DI. Intracoronary optical coherence tomography: a comprehensive review clinical and research applications. JACC Cardiovasc Interv. 2009 Nov;2(11):1035-46. doi: 10.1016/j.jcin.2009.06.019. PMID 19926041
- [Background] Kubo T, Imanishi T, Kashiwagi M, Ikejima H, Tsujioka H, Kuroi A, Ishibashi K, Komukai K, Tanimoto T, Ino Y, Kitabata H, Takarada S, Tanaka A, Mizukoshi M, Akasaka T. Multiple coronary lesion instability in patients with acute myocardial infarction as determined by optical coherence tomography. Am J Cardiol. 2010 Feb 1;105(3):318-22. doi: 10.1016/j.amjcard.2009.09.032. Epub 2009 Dec 22. PMID 20102942
- [Background] Kubo T, Imanishi T, Takarada S, Kuroi A, Ueno S, Yamano T, Tanimoto T, Matsuo Y, Masho T, Kitabata H, Tsuda K, Tomobuchi Y, Akasaka T. Assessment of culprit lesion morphology in acute myocardial infarction: ability of optical coherence tomography compared with intravascular ultrasound and coronary angioscopy. J Am Coll Cardiol. 2007 Sep 4;50(10):933-9. doi: 10.1016/j.jacc.2007.04.082. Epub 2007 Aug 20. PMID 17765119